CLINICAL TRIAL: NCT04495270
Title: Two-year Treatment Outcomes of Teeth With Apical Periodontitis Based on Cone-beam Computed Tomography and Estimated by Means of Periapical and Endodontic Status Scale
Brief Title: 2-year Treatment Outcomes of Teeth Estimated by Means of Periapical and Endodontic Status Scale
Status: Completed | Type: Observational
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Jelena Gudac, Principal Investigator, Lithuanian University of Health Sciences
Other Study IDs: BE-2-27
Record Dates: First submitted 2020-07-22; First posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Periapical Periodontitis; Treatment Outcome
Keywords: Cone-beam computed tomography; Periapical periodontitis; Scale; Treatment outcome
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinical observation: All study patients were examined by 1 endodontist clinically and radiographically at baseline and after follow up of endodontic treatment.
  Interventions: Diagnostic Test: Analysis of treatment outcomes of teeth with apical periodontitis based on cone-beam computed tomography and estimated by means of Periapical and Endodontic Status Scale"

INTERVENTIONS:
Diagnostic Test: Analysis of treatment outcomes of teeth with apical periodontitis based on cone-beam computed tomography and estimated by means of Periapical and Endodontic Status Scale" — Patients were examined by cone-beam computed tomography at baseline and in 24 months after endodontic treatment. Treatment outcome was evaluated using estimates of periapical radiolucencies in size, relation with anatomical structures and location.

SUMMARY:
Objectives: Evaluation of endodontic treatment success is largely based on radiographical assessment of anatomical and treatment-related parameters of teeth with apical periodontitis (AP). This study aimed to analyse 2-year treatment outcomes of teeth with AP based on radiographical changes, and to evaluate prognostic validity of Periapical and Endodontic Status Scale (PESS).

Materials and Methods: 128 patients (176 teeth) were examined by cone-beam computed tomography at baseline and in 24 months after endodontic treatment. Treatment outcome was evaluated using estimates of periapical radiolucencies in size, relation with anatomical structures and location. Strength of associations between these and treatment-related parameters was tested by logistic regression analysis. Predictive validity of PESS was verified by estimating association between treatment risk groups defined at baseline and negative outcome.

DETAILED DESCRIPTION:
Study sample The study participants were adult patients, admitted for general oral rehabilitation to Vilnius Implantology Center, Lithuania, and referred for treatment to a specialist in endodontics during the period December 2016 - December 2019. A total of 140 patients, with 200 teeth with AP, were invited to participate in the study. Ten patients were excluded according to the inclusion criteria, and 2 patients declined to participate. Finally, 128 patients with 176 teeth with AP, agreed to participate in this study. The mean age of the participants was 46 years, range 18-70 years, (SD =12.3).

The inclusion criteria were as follows:

* no systemic diseases present;
* at least one tooth with the diagnosis of AP (necrotic pulp and/or filled root canals) present;
* sufficient periodontal support (absence of clinical periodontal inflammation on an anatomically intact or, on a reduced periodontium of the teeth indicated for treatment);
* baseline CBCT images available (performed for general oral rehabilitation planning purposes, no earlier than one month prior to endodontic procedures).

The diagnosis of apical periodontitis was based on the clinical tests of pulp vitality (sensitivity to heat and cold), percussion, palpation, presence of abnormal bite, swelling, caries, sinus tracts, of unstimulated/stimulated pain, and on the radiological findings. A total of 176 teeth (403 root canals) were subjected to endodontic treatment.

Pregnant women, immunosuppressed patients, and patients presenting with un-restorable teeth (e.g., deep root caries lesion, coronal cracks, root fracture) or, with the probing depths >5 mm around the marginal bone were excluded.

All the participants gave written informed consent to be involved in the clinical trial. The study protocol was approved by the Ethical Committee of Biomedical studies, Lithuania (Protocol No 111; 10.03.2016; edition No BE-2-27; 20.12.2016).

Clinical and radiographic examinations:

All study patients were examined clinically and radiographically at baseline, and in 24 months (further on, referred as "2 years") after endodontic treatment. The intermediate follow-up examinations were set at 12 months' time point, however, only the final study results are discussed in the present report.

The clinical examinations were performed by one examiner (JG) and included standard tests such as percussion, palpation, evaluation of coronal seal, of tooth mobility and of the periodontal probing depth. All diagnostic procedures were performed in a dental chair using a dental mirror and explorer (Dentsply Maillefer, Ballaigues, Switzerland). The case history (presence of clinical symptoms, complaints, the time of the previous treatment) was obtained from every patient.

Radiographical examinations of the patients were performed with CBCT imaging, and with digital radiography. For the present study purposes, only CBCT data were included in the analysis. The baseline CBCT images were already available following the general diagnostic and treatment plan. The follow-up CBCT was performed in 2 years after the endodontic treatment, only for the respective maxillary or mandibular arch. All images were made with i-CAT scanner (Imaging Sciences International Inc., Hatfield, PA, USA), the exposure parameters were as follows: 84 kV, 5 mA, 0.3 mm voxel resolution, 6x16 and 6x6 cm field of view, 18.3s and 5s acquisition time at baseline and at the final examination, respectively. The CBCT images were viewed as an original i-Cat presentation (Apple, Cupertino, CA, USA) on the computers with a 27-inch flat panel display with a pixel resolution of 2.560 x 1.440 with dimmed ambient light, less than 50 lux, without time restrictions. A total of 256 (128 baseline and 128 follow up) CBCT images were coded and analyzed by the same examiner (JG), without knowledge of the clinical data.

The radiographical assessment of the periapical status of the teeth was performed following the Periapical and Endodontic Status Scale (PESS).

ELIGIBILITY:
Inclusion Criteria:

* no systemic diseases present;
* at least one tooth with the diagnosis of AP (necrotic pulp and/or filled root canals) present;
* sufficient periodontal support (absence of clinical periodontal inflammation on an anatomically intact or, on a reduced periodontium [13] of the teeth indicated for treatment);
* baseline CBCT images available (performed for general oral rehabilitation planning purposes, no earlier than one month prior to endodontic procedures).

Exclusion Criteria:

* Pregnant women;
* immunosuppressed patient
* patients presenting with un-restorable teeth (e.g., deep root caries lesion, coronal cracks, root fracture)
* with the probing depths >5 mm around the marginal bone.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study participants were adult patients, admitted for general oral rehabilitation and referred for treatment to a specialist in endodontics
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
The positive treatment outcome | 24 months
  Decreased periapical radiolucency, with respect to it's size, or/and relation with anatomical structures, location (respective parameters S, R, and D). Moreover, the unchanged mild severity scores S1, D1, and R1 were regarded as positive outcome as well. The minimum value 0 (means better outcome), the maximum value - 3 (means worse outcome).
The negative treatment outcome | 24 months
  Increased/unchanged periapical radiolucency in size, or/and in relation with anatomical structures, or/and in location (respective parameters S, R, and D). By comparing the baseline and the final CBCT images all transition events from the lower to the higher scores and the following unchanged scores were considered as negative treatment outcomes.The minimum value 0 (means better outcome), the maximum value - 3 (means worse outcome).

IPD SHARING:
Plan to Share IPD: No